CLINICAL TRIAL: NCT04697810
Title: A Phase 2B Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Namodenoson in the Treatment of Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Namodenoson in the Treatment of Non-Alcoholic Steatohepatitis (NASH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF102-212LD
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-chloro-N(6)-(3-iodobenzyl)adenosine-5'-N-methyluronamide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 2:1 ratio of namodenoson 25 mg or matching placebo, according to a computer-generated randomization schedule. Blocked randomization will be programmed using a pre-specified block size. Double-blinding will be maintained throughout the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo capsules are identical in appearance to namodenoson capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Namodenoson (Experimental): Namodenoson capsules orally 25 mg every 12 hours for 36 weeks
  Interventions: Drug: Namodenoson
- Placebo (Placebo Comparator): Matching placebo capsules orally 25 mg every 12 hours for 36 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Namodenoson — 25 mg q12hours x 36 weeks
  Other Names: CF102
  Arms: Namodenoson
Drug: Placebo — Matching capsules q12hours x 36 weeks
  Other Names: Inactive control
  Arms: Placebo

SUMMARY:
Subjects with biopsy-proven NASH will be randomly assigned in a 2:1 ratio to oral doses of namodenoson 25 mg every 12 hours or matching placebo every 12 hours for 36 weeks. Subjects will be evaluated regularly for safety, and efficacy biomarkers will be measured at Baseline and Weeks 6, 12, 24, and 36. At Week 36, all subjects will undergo liver biopsy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study in subjects with a diagnosis of NASH and F1-3 fibrosis. Subjects will undergo Screening procedures during the 6 weeks preceding Baseline. Subjects (n = ~114) will be randomly assigned in a 2:1 ratio to oral doses of namodenoson 25 mg every 12 hours or matching placebo every 12 hours for 36 weeks. Subjects will be evaluated regularly for safety, and efficacy biomarkers will be measured at Baseline and Weeks 6, 12, 24, and 36. At Week 36, all subjects will undergo post-treatment liver biopsy, which will be interpreted by a blinded expert hepatopathologist. Subjects will return for a follow-up visit 6 weeks after completion of the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. AST at Screening of ≥20 IU/L.
3. FibroScan LSM ≥8.5 kPa
4. Diagnosis of NASH by biopsy at Screening showing NAS ≥4 by central read, with a score of at least 1 point in each of the 3 histologic categories of steatosis, inflammation, and hepatocellular ballooning (Kleiner 2005). If the subject has had a qualifying liver biopsy within 6 months prior to Baseline and the slides are available for central read prior to randomization, this biopsy can be waived.
5. Concomitant biopsy-proven Stage 1-3 hepatic fibrosis by NASH CRN criteria by central read (Kleiner 2005).
6. At least 2 of the following criteria for the metabolic syndrome:

   * Obesity, defined waist circumference >88 cm for women or >102 cm for men
   * Hypertriglyceridemia, defined as >150 mg/dL (>1.7 mmol/L) or on drug treatment for hypertriglyceridemia
   * Reduced high-density lipoprotein (HDL) cholesterol, defined as <40 mg/dL (<1.03 mmol/L) in men or <50 mg/dL (<1.3 mmol/L) in women
   * History of hypertension, currently controlled in the judgment of the Investigator
   * Elevated fasting glucose, defined as ≥100 mg/dL (≥5.6 mmol/L).
7. Acceptable hepatic metabolic and synthetic function, as indicated at Screening by:

   * Serum albumin ≥3.5 gm/dL
   * International normalized ratio ≤1.3
   * Serum total bilirubin ≤2.0 mg/dL (unless subject has known Gilbert's Syndrome).
8. The following laboratory values must be documented at Screening:

   * Absolute neutrophil count at least 1.0 x 109/L
   * Platelet count at least 150 x 109/L
   * Estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m2
9. Female subjects may be enrolled if they are not of childbearing potential, permanently sterile or are post-menopausal, defined as no menses for at least 1 year without an alternative medical cause and FSH levels in the post-menopausal range.
10. Male subjects must refrain from sperm donation during treatment and until at least 90 days after the end of study drug dosing. Male subjects with fertile or pregnant partners must agree to use condoms throughout the course of the trial and for 3 months after.
11. Patients taking herbal supplements, homeopathic medications, or other alternative treatments, must be on a stable regimen for at least 3 months prior to randomization.
12. Understand and provide written informed consent to participate.
13. Willing to undergo 2 liver biopsies.
14. Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other study-related procedures.

Exclusion Criteria:

1. Ascites, hepatic encephalopathy, or other clinical evidence of cirrhosis.
2. Other active acute or chronic liver disease, such as autoimmune hepatitis, hepatitis B, hepatitis C, alcoholic liver disease, or hepatocellular carcinoma.
3. Seropositivity for markers of viral hepatitis or human immunodeficiency virus (HIV) at Screening.
4. Weight loss of >5% within 3 months prior to Baseline.
5. History of bariatric surgery within 5 years of Screening.
6. Diabetes mellitus other than Type II.
7. Hemoglobin A1c >9.0% (subjects with diabetes).
8. Any contraindication to percutaneous liver biopsy.
9. Daily alcohol intake >20 g (2 units)/day for women and 30 g (3 units)/day for men (on average), as per Alcohol Use Disorders Identification Test (AUDIT) questionnaire.
10. Treatment with therapeutic doses of Vitamin E (≥800-1000 IU daily), or any of the following anti-diabetic medications: GLP-1 receptor agonists (such as Januvia [sitagliptin], Byetta [incretin], etc.), pioglitazone, or SGLT2 inhibitors ("gliflozin" drugs); unless the dose and regimen has been stable for at least 3 months.
11. Active rheumatoid arthritis treated with small-molecule (including methotrexate) or biologic disease-modifying anti-rheumatic agent concurrently or within 1 year.
12. Use of any immunosuppressive medication, anti-inflammatory monoclonal antibody treatment, or chronic systemic corticosteroids >10 mg prednisone-equivalent concurrently or within 1 year.
13. More than 7 days of treatment with valproic acid, tamoxifen, amiodarone, or anti-cholinergic agents within 3 months.
14. Uncontrolled or clinically unstable thyroid disease.
15. Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4), or other heart disease which is, in the Investigator's judgment, clinically unstable.
16. Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months.
17. QTcF interval on Screening Visit ECG or an average of triplicate Baseline Visit ECGs > 450 milliseconds (msec) for males or > 470 msec for females.
18. A condition which increases proarrhythmic risk, including hypokalemia, hypomagnesemia, or congenital Long QT Syndrome.
19. Ongoing or planned use of a concomitant medication that is on the CredibleMedsTM list of drugs known to cause Torsades des Pointes.
20. Active gastrointestinal disease which could interfere with the absorption of oral medication.
21. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Non-Alcoholic Fatty Liver Disease (NAFLD) activity score (NAS) | 36 weeks
  Proportion of subjects who achieve a ≥2-point improvement in the non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of the Non-Alcoholic Steatohepatitis Clinical Research Network (NASH CRN)
Adverse events (AEs) | 36 weeks
  Incidence of AEs

SECONDARY OUTCOMES:
Alanine transaminase (ALT) mean | 36 weeks
  Mean percent change from Baseline in serum ALT level
Steady-state blood level of namodenoson | 36 weeks
  Plasma trough concentration (ng/mL) of namodenoson taken at pre-dose samples

OTHER OUTCOMES:
ALT absolute | 36 weeks
  Absolute change from Baseline in serum ALT
ALT threshold | 36 weeks
  Proportion of subjects who achieve ≥17-point reduction from Baseline in serum ALT
Weight | 36 weeks
  Change from Baseline in body weight
Adiponectin | 36 weeks
  Change from Baseline in serum adiponectin level
Released N-terminal pro-peptide of type III collagen neoepitope (Pro-C3) | 36 weeks
  Change from Baseline in Pro-C3
Serum Enhanced Liver Fibrosis (ELF) Score | 36 weeks
  Change from Baseline in ELF Score, which is a continuous scale starting at zero, with higher scores indicating more severe disease
FibroScan controlled attenuation parameter (CAP) | 36 weeks
  Change from Baseline in CAP
FibroScan-AST (FAST) Score | 36 weeks
  Change from Baseline in FAST Score, which is a decimal score from 0 to 1, with higher scores indicating more severe disease
Aspartate transaminase (AST) | 36 weeks
  Change from Baseline in serum AST
Gamma-glutamyl transferase (GGT) | 36 weeks
  Change from Baseline in serum GGT
Fibrosis-4 (Fib-4) Index | 36 weeks
  Change from Baseline in Fib-4 Index
NASH resolution | 36 weeks
  Proportion of subjects who achieve histologic NASH resolution as defined by a ballooning score of 0 and an inflammation score of 0-1 without worsening of fibrosis
NASH fibrosis improvement | 36 weeks
  Proportion of subjects who achieve histologic NASH improvement by at least 1 point without worsening of NASH

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — BioStrategics Consulting Ltd
Locations (24):
- Bosnia and Herzegovina (2):
  - 941 Univ of Clinical Centre of the Republic of Srpska, Banja Luka
  - 942 Health Inst General Hospital, Dept of Internal Medicine, Prijedor
- Bulgaria (8):
  - 934 Second Dept of Internal Disease, MHAT Sveta Karidad EAD, Plovdiv
  - 932 Office of Gastroenterology, Medical Center Sansi EOOD, Rousse
  - 931 Clinic of Gastroenterology, Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia, Sofia
  - 933 Clinic of Gastroenterology, University Multiprofile Hosptial for Active Treatment, Sofia
  - 935 Dept of Gastroent., Univ Multiprofile Hospital for Active Treatment and Emergency Medicine, Sofia
  - 936 Office of Gastroenterology, Diagnostic - Consultative Center XX, Sofia
  - 937 Office of Gastroenterology, Diagnostic - Consultative Center Alexandrovska, Sofia
  - 938 Clinic of Gastroenterology, University Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski", Sofia
- Israel (2):
  - 517 Saroka University Medical Center, Beersheba
  - Hadassah Medical Center, Jerusalem
- Moldova (2):
  - 911 IMSP Spitalul Clinic Republican "Timofei Mosneaga", Chisinau
  - 912 SP Spitalul Ministerului Sanatatii, Muncii si Protectiei Sociale, Chisinau
- Romania (6):
  - 903 Central Pentru Studiul Metabolismului, Bucharest
  - 904 SUUMC Carol Davilla, Department Diabet, Bucharest
  - 906 Spitalul Sfanta Maria, Bucharest
  - 902 Cluj County Clinical Emergency Hospital, 3rd Dept of Internal Medicine, Cluj-Napoca
  - 901 Medical Center Dr. Ianosi, Craiova
  - 905 County Hospital Timisoara, Timișoara
- Serbia (4):
  - 922 UCC Zvezdara Belgrade, Belgrade
  - 923 Military Medical Academy Belgrade, Belgrade
  - 924 CHC "dr Dragisa Misovic" - Dedinje Belgrade, Belgrade
  - 921 UCC Nis, Niš

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen S, Stemmer SM, Zozulya G, Ochaion A, Patoka R, Barer F, Bar-Yehuda S, Rath-Wolfson L, Jacobson KA, Fishman P. CF102 an A3 adenosine receptor agonist mediates anti-tumor and anti-inflammatory effects in the liver. J Cell Physiol. 2011 Sep;226(9):2438-47. doi: 10.1002/jcp.22593. PMID 21660967
- [Background] Safadi R, Braun M, Francis A, Milgrom Y, Massarwa M, Hakimian D, Hazou W, Issachar A, Harpaz Z, Farbstein M, Itzhak I, Lev-Cohain N, Bareket-Samish A, Silverman MH, Fishman P. Randomised clinical trial: A phase 2 double-blind study of namodenoson in non-alcoholic fatty liver disease and steatohepatitis. Aliment Pharmacol Ther. 2021 Dec;54(11-12):1405-1415. doi: 10.1111/apt.16664. Epub 2021 Oct 20. PMID 34671996
- See also: Sponsor website — https://www.canfite.com/